CLINICAL TRIAL: NCT05894720
Title: Effect of Thrower's Ten Exercises on Flick Movement Kinematics in Underwater Hockey
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Leyla Eraslan, Assistant Professor, Hacettepe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GO 13/307
Record Dates: First submitted 2023-05-29; First posted 2023-06-08 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Hockey
Keywords: underwater hockey; kinematics; throwers ten exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Thrower's Ten Exercise Group (Experimental): the athletes were subjected to "Thrower's Ten" exercise program under the supervision of the same physiotherapist 3 days a week for a period of 6 weeks in addition to the routine practice programs thereof. Each session started with a 10-minute warm-up program and ended with a 10-minute cool-down program. The warm-up program included low-intensity aerobic activities and short stretching exercises. Stretching exercises for anterior-posterior-inferior capsule, right and left trapezoid muscles, chintug as well as posterior-lateral neck and latissimus dorsi muscles were given. Following the exercises, the athletes were made to perform low-intensity jogging and static stretching exercises. All athletes, who were included in the study sample, continued attending their 2-hour routine pool practice on 4 days a week in addition to the "Thrower's Ten" exercises for 6 weeks.
  Interventions: Other: Thrower's Ten Exercise Group

INTERVENTIONS:
Other: Thrower's Ten Exercise Group — the athletes were subjected to "Thrower's Ten" exercise program under the supervision of the same physiotherapist 3 days a week for a period of 6 weeks in addition to their routine practice programs.

SUMMARY:
Underwater hockey is a team game which is played at the bottom of the swimming pool with palettes, a mask, a snorkel, earmuffs, a stick, and a puck. The aim of the game is for one of the teams to try to score goals to the goalpost of the other by using a flicking movement. The players can drag the puck, being a kind of ball, or pass it to a teammate to reach the opponent's goalpost. The puck is passed by way of pushing or flicking.

The Thrower's Ten exercises are used for such sports branches, which involve the upper extremity and particularly the overhead activity and throwing, in order to ensure coordination, proprioception, balance and symmetry in the double upper extremity. The Thrower's Ten exercises are comprised of special exercises selected for the improvement of the flexibility, strength and endurance of the major muscles that are frequently used for throwing and overhead activity such as deltoid muscles, supraspinatus muscles, latissimus dorsi, biceps, triceps and wrist extensors. The Thrower's Ten exercises are an exercise program that focuses on the scapular muscles, particularly on posterior rotator cuff muscles in order to ensure the balance of the anterior and the posterior shoulder muscles.

The aim of this study is to evaluate the effects of The Thrower's Ten exercise program on the flicking movements in underwater hockey players.

DETAILED DESCRIPTION:
Underwater hockey is a team game which is played at the bottom of the swimming pool with palettes, a mask, a snorkel, earmuffs, a stick, and a puck. The aim of the game is for one of the teams to try to score goals to the goalpost of the other by using a flicking movement. The players can drag the puck, being a kind of ball, or pass it to a teammate to reach the opponent's goalpost. The puck is passed by way of pushing or flicking.

The Thrower's Ten exercises are used for such sports branches, which involve the upper extremity and particularly the overhead activity and throwing, in order to ensure coordination, proprioception, balance and symmetry in the double upper extremity. The Thrower's Ten exercises are comprised of special exercises selected for the improvement of the flexibility, strength and endurance of the major muscles that are frequently used for throwing and overhead activity such as deltoid muscles, supraspinatus muscles, latissimus dorsi, biceps, triceps and wrist extensors. The Thrower's Ten exercises are an exercise program that focuses on the scapular muscles, particularly on posterior rotator cuff muscles in order to ensure the balance of the anterior and the posterior shoulder muscles.

The aim of this study is to evaluate the effects of The Thrower's Ten exercise program on the flicking movements in underwater hockey players.

ELIGIBILITY:
Inclusion Criteria:

* 1st league healthy underwater hockey players

Exclusion Criteria:

* Previous shoulder injury

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Flicking Distance Measurement | from baseline to six weeks after treatment sessions
  Flicking Distance will be measured by using video cameras. Assessment will be recorded at baseline and the end of the six weeks treatment sessions

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Faculty of Health Sciences, Dept. of Physiotherapy and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
We will share IPD when we recruiting the patients